CLINICAL TRIAL: NCT06001177
Title: A Phase 2a Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of KAN-101 In Participants With Celiac Disease
Brief Title: A Study of Efficacy, Safety, and Tolerability of KAN-101 in People With Celiac Disease
Acronym: SynCeD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanyos Bio, Inc., a wholly-owned subsidiary of Anokion SA (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Anokion SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAN-101-03
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Celiac Disease; Coeliac Disease
Keywords: celiac disease; HLA-DQ2.5; gluten free diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, placebo-controlled study with approximately 52 participants that will receive KAN-101 or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants and their caregivers, investigators and other staff, and sponsor staff involved in the study team will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): All eligible participants will receive 3 intravenous (IV) infusions of KAN-101
  Interventions: Drug: KAN-101
- Group 2 (Placebo Comparator): All eligible participants will receive 3 intravenous (IV) infusions of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAN-101 — Dose KAN-101 Intravenous (IV) Infusion
  Other Names: Group 1, Treatment Arm
  Arms: Group 1
Drug: Placebo — Placebo Intravenous (IV) Infusion
  Other Names: Group 2, Placebo Comparator Arm
  Arms: Group 2

SUMMARY:
The study goal is to evaluate the efficacy, safety, and tolerability of KAN-101 in participants with Celiac Disease (CeD)

DETAILED DESCRIPTION:
Study KAN-101-03 is a multi-center, double-blind, placebo-controlled Phase 2a study to examine whether KAN-101 confers protection from gluten exposure induced histological changes in the duodenum and to further evaluate the safety/tolerability of KAN-101 in adult participants (≥18 years) with CeD on a gluten free diet. Approximately 52 participants who meet study inclusion/exclusion criteria will be randomized 1:1 to receive KAN-101 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of celiac disease based on histology and positive celiac serology
* HLA-DQ2.5 genotype
* Gluten-free diet for at least 12 months
* Negative or weak positive for transglutaminase IgA and negative or weak positive for DGP-IgA/IgG during screening
* Screening intestinal biopsy demonstrating Vh:Cd ratio of 2.3 or higher

Exclusion Criteria:

* Refractory celiac disease
* HLA-DQ8 genotype
* Selective IgA deficiency
* Diagnosis of type-I diabetes
* Other Active gastrointestinal diseases
* History of dermatitis herpetiformis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Anokion SA
Locations (28):
- United States (6):
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Unlimited Medical Research Group, Hialeah Gardens, Florida
  - Homestead Associates in Research Inc., Miami, Florida
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Canada (5):
  - McMaster University, Hamilton, Ontario
  - LHSC, London, Ontario
  - Centre Intégré de Santé et de Services Sociaux-Chaudière Appalaches - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Hopital Du Sacre-Coeur De Montreal, Montreal, Quebec
  - Diex Recherche Quebec Inc., Québec, Quebec
- Finland (3):
  - Tays Research Services, Tampere, Pirkanmaa
  - Clinical Research Services Turku, Turku, Southwest Finland
  - CRST Helsinki Oy, Helsinki, Uusimaa
- Studiengesellschaft BSF Unternehmergesellschaft, Halle, Saxony-Anhalt, Germany
- Ireland (3):
  - Connolly Hospital, Dublin, Dublin
  - Our Lady of Lourdes Hospital, Drogheda, Louth
  - Midland Regional Hospital Mullingar, Mullingar, Westmeath
- Israel (4):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
- Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht, South Holland, Netherlands
- Poland (5):
  - Gastromed Sp. z o. o., Torun, Kuyavian-Pomeranian Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
  - MZ Badania Slowik Zymla Spolka Jawna, Knurów, Silesian Voivodeship
  - Centrum Medyczne Med-Gastr Sp. z o.o., Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray JA, Wassaf D, Dunn K, Arora S, Winkle P, Stacey H, Cooper S, Goldstein KE, Manchanda R, Kontos S, Grebe KM. Safety and tolerability of KAN-101, a liver-targeted immune tolerance therapy, in patients with coeliac disease (ACeD): a phase 1 trial. Lancet Gastroenterol Hepatol. 2023 Aug;8(8):735-747. doi: 10.1016/S2468-1253(23)00107-3. Epub 2023 Jun 14. PMID 37329900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 participants were enrolled and treated, of which 50 participants completed the study, 2 participants discontinued from the treatment phase, and 3 participants discontinued from the observation phase.
Groups:
- 0.6 mg/kg KAN-101: All enrolled participants received 0.6 mg/kg of KAN-101 via intravenous (IV) infusions every 3 days starting on Day 1 and ending on Day 7
  KAN-101: 0.6 mg/kg KAN-101 Intravenous (IV) Infusion
- Placebo: All enrolled participants received intravenous (IV) infusions of placebo every 3 days starting on Day 1 and ending on Day 7
  Placebo: Placebo Intravenous (IV) Infusion
Period: Treatment Phase
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Started | 28 | 27
Completed | 26 | 27
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Observation Phase
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Started | 26 | 27
Completed | 25 | 25
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow-Up
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.6 mg/kg KAN-101 | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (15.10) | 39.7 (13.96) | 39.3 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 28 | 24 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 167.76 (9.055) | 165.64 (8.635) | 166.72 (8.834)
Weight [Mean (Standard Deviation); unit: kg] | 71.30 (16.183) | 71.23 (13.386) | 71.26 (14.738)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.30 (5.290) | 26.07 (5.191) | 25.68 (5.207)
Time since First CeD Diagnosis [Mean (Standard Deviation); unit: years] | 7.8 (5.36) | 9.4 (5.57) | 8.6 (5.48)
Time on Gluten-Free Diet (GFD) [Mean (Standard Deviation); unit: years] | 7.4 (5.34) | 7.5 (5.66) | 7.5 (5.45)
Human Leukocyte Antigen (HLA) Genotype [Number; unit: participants]
  Positive | 27 | 27 | 54
  Negative | 1 | 0 | 1
Positive Celiac Serology at Diagnosis [Number; unit: participants]
  TISSUE TRANSGLUTAMINASE IGA ANTIBODY (TTG-IGA) | 26 | 25 | 51
  TISSUE TRANSGLUTAMINASE IGG ANTIBODY (TTG-IGG) | 5 | 1 | 6
  DEAMIDATED GLIADIN PEPTIDE IGA (DGP-IGA) | 3 | 0 | 3
  DEAMIDATED GLIADIN PEPTIDE IGG (DGP-IGG) | 4 | 1 | 5
Positive Histology at Diagnosis [Number; unit: participants] — Marsh 0: Normal intestinal villi with no signs of damage. Marsh 1: Increased intraepithelial lymphocytes, but no villous atrophy. Marsh 2: Increased intraepithelial lymphocytes and crypt hyperplasia. Marsh 3: The classic spectrum for celiac disease, with increased lymphocytes, crypt hyperplasia, and villous atrophy.
  3a: Mild villous atrophy. 3b: Marked villous atrophy. 3c: Total villous atrophy, or complete flattening of the villi. Marsh 4: Total villous atrophy with shrunken crypts.
  participants
    EVIDENCE OF VILLOUS ATROPHY (NO MARSH SCORE REPORTED) | 18 | 16 | 34
    MARSH SCORE 2 | 0 | 3 | 3
    MARSH SCORE 3A | 4 | 1 | 5
    MARSH SCORE 3B | 3 | 5 | 8
    MARSH SCORE 3C | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Villous Height to Crypt Depth (Vh:Cd) as Assessed by Esophagogastroduodenoscopy With Biopsy After 2-week Gluten Challenge (GC)
Description: KAN-101 attenuated GC-induced changes in duodenal histology as measured by the Vh:Cd ratio.
Time Frame: Baseline and Day 29
Population: Full Analysis Set - All participants who were randomly assigned to the study intervention, received all 3 doses of the study intervention, and completed at least 7 days of the 2-week GC without prohibited medications. Participants were analyzed according to the study intervention they were randomized.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Number analyzed (Participants) | 25 | 25
ratio | -0.85 (0.707) | -0.61 (0.614)
Statistical Analysis 1: Comparison: 0.6 mg/kg KAN-101 vs Placebo; Test type: Superiority; p = 0.1668, ANCOVA — P-value was based on an ANCOVA model with treatment as a factor and baseline as a covariate; Least Squares Mean Difference = -0.26, 95% CI 2-sided [-0.63 to 0.11], Standard Error of Mean 0.185

2. Secondary Outcome: Change in Magnitude of Interleukin-2 (IL-2) Response From Day 15 (First Day of GC) Pre-GC to Day 15 Post GC
Time Frame: From Day 15 pre-GC to Day 15 post GC
Population: Biomarker Analysis Set - All participants who were randomly assigned to the study intervention, received any portion of the study intervention, and had completed the GC on Day 15 without prohibited medications. Participants were analyzed according to the study intervention they were randomized.
Measure: Mean (Standard Deviation); unit: international unit
Groups:
- Placebo: All enrolled participants received intravenous (IV) infusions every 3 days of placebo starting on Day 1 and ending on Day 7
  Placebo: Placebo Intravenous (IV) Infusion
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Number analyzed (Participants) | 26 | 27
international unit | 31.8 (95.86) | 31.1 (102.30)

3. Secondary Outcome: Changes From Baseline in Intraepithelial Lymphocyte (IEL) Density in Duodenum Biopsy After 2-week GC
Time Frame: Baseline and Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: cells per 100 epithelial cells
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Number analyzed (Participants) | 25 | 25
cells per 100 epithelial cells | 20.68 (17.447) | 17.36 (16.286)

4. Secondary Outcome: Incidence and Severity of Treatment Emergent Adverse Events (TEAE) as Assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious adverse events. SAE was defined as any untoward medical occurrence that, at any dose resulted in any of the following outcomes: death; life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or that was considered as an important medical event. According to NCI CTCAE version 5: Grade 1= mild AE; Grade 2= moderate AE; Grade 3=severe AE; Grade 4= life-threatening consequences and urgent intervention indicated; Grade 5= death related to AE. An AE was considered treatment-emergent relative to a given treatment if the event start date is during the on-treatment period (including on the date of first dose).
Time Frame: From the time the participant provided informed consent through Day 42.
Population: Safety Analysis Set - All participants who received any portion of the study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Number analyzed (Participants) | 28 | 27
Participants
  TEAE | 25 | 22
  SAE | 1 | 0
  Grade 2 TEAE | 0 | 1
  Grade 3 or higher TEAE | 1 | 0

5. Secondary Outcome: Incidence by Visit of KAN-101 Antidrug Antibody (ADA)
Time Frame: Up to 42 days
Population: Safety analysis set - all participants who received any portion of study intervention. Participants with at least 1 positive response post-treatment.
Measure: Number; unit: participants
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
Number analyzed (Participants) | 28 | 0
participants
  Baseline | 0 |
  Day 7: number analyzed (Participants) | 27 | 0
  Day 7 | 0 |
  Day 29: number analyzed (Participants) | 24 | 0
  Day 29 | 3 |
  Day 42: number analyzed (Participants) | 25 | 0
  Day 42 | 5 |

6. Secondary Outcome: KAN-101 Plasma Concentration: AUCinf
Description: Area under the plasma-concentration time curve from time 0 extrapolated to infinite time.
Time Frame: 0 minutes, 30 minutes, 2 hours 30 minutes, 4 hours post dose on day 1 and day 7
Population: AUC could not be determined due to limited data points. Samples at the terminal elimination phase were below limit of quantification.
Measure: Mean (Standard Deviation); unit: hr/mL
Arm/Group | 0.6 mg/kg KAN-101
Number analyzed (Participants) | 28
hr/mL | NA — AUC could not be determined due to limited data points. Samples at the terminal elimination phase were below limit of quantification.

7. Secondary Outcome: KAN-101 Plasma Concentration: AUClast
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast).
Time Frame: 0 minutes, 30 minutes, 2 hours 30 minutes, 4 hours post dose on day 1 and day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr/mL
Arm/Group | 0.6 mg/kg KAN-101
Number analyzed (Participants) | 28
hr/mL | NA — AUC could not be determined due to limited data points. Samples at the terminal elimination phase were below limit of quantification.

8. Secondary Outcome: KAN-101 Plasma Concentration: Cmax
Description: Maximum plasma concentration.
Time Frame: 0 minutes, 30 minutes, 2 hours 30 minutes, 4 hours post dose on day 1 and day 7
Population: PK Analysis Set - All participants who receive any portion of study intervention and have at least one post-dose concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.6 mg/kg KAN-101
Number analyzed (Participants) | 28
ng/mL
  Day 1: number analyzed (Participants) | 27
  Day 1 | 3141.9 (39)
  Day 7: number analyzed (Participants) | 26
  Day 7 | 4107.9 (66.7)

9. Secondary Outcome: KAN-101 Plasma Concentration: Tmax
Description: Time to reach Cmax.
Time Frame: 0 minutes, 30 minutes, 2 hours 30 minutes, 4 hours post dose on day 1 and day 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.6 mg/kg KAN-101
Number analyzed (Participants) | 28
h
  Day 1: number analyzed (Participants) | 27
  Day 1 | 0.7 (0.48)
  Day 7: number analyzed (Participants) | 26
  Day 7 | 0.6 (0.13)

10. Secondary Outcome: KAN-101 Plasma Concentration: T1/2
Description: Terminal phase half-life.
Time Frame: 0 minutes, 30 minutes, 2 hours 30 minutes, 4 hours post dose on day 1 and day 7
Population: T1/2 could not be determined due to limited data points. Samples at the terminal elimination phase were below limit of quantification.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 0.6 mg/kg KAN-101
Number analyzed (Participants) | 28
hour | NA — T1/2 could not be determined due to limited data points. Samples at the terminal elimination phase were below limit of quantification.

ADVERSE EVENTS:
Time Frame: From the time the participant provided informed consent through Day 42.
Arm/Group | 0.6 mg/kg KAN-101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27
Other Adverse Events (participants affected / at risk) | 24/28 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg/kg KAN-101 (N=28) | Placebo (N=27)
Fracture treatment (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg/kg KAN-101 (N=28) | Placebo (N=27)
Vertigo (Ear and labyrinth disorders) | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 7 | 8
Abdominal pain (Gastrointestinal disorders) | 11 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 9
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Eructation (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 16 | 11
Vomiting (Gastrointestinal disorders) | 9 | 4
Fatigue (General disorders) | 8 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Brain fog (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 6 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT06001177/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT06001177/SAP_001.pdf